CLINICAL TRIAL: NCT07337850
Title: FAP 2: Utility of Gallium-68-Fibroblast Activation Protein Inhibitor (FAPI) PET in Biliary Tract Cancers: A Prospective Study
Brief Title: Prospective Evaluation of 68Ga-FAPI PET in Biliary Cancers
Acronym: FAPi-2
Status: Recruiting | Type: Observational
Sponsor: Tata Memorial Centre (Other)
Responsible Party: Sponsor
Other Study IDs: Study no:- 4455; 6429 (Other Grant/Funding Number: Tata Memorial Hospital)
Record Dates: First submitted 2026-01-01; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Gall Bladder Cancer; Intrahepatic Cholangiocarcinoma (Icc)
Keywords: FAPI PET/CT; Gallium-68 FAPI; Biliary Tract Cancer; Gallbladder Cancer; Cholangiocarcinoma; Intrahepatic Cholangiocarcinoma (iHCC)
MeSH Terms: conditions — Gallbladder Neoplasms; Cholangiocarcinoma; Cirrhosis, Familial, with Pulmonary Hypertension; Biliary Tract Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: gallium-68-Fibroblast Activation Protein Inhibitor — Gallium-68 Fibroblast Activation Protein Inhibitor (Ga-68 FAPI) is a radiolabeled molecular imaging tracer used for PET/CT imaging. It targets Fibroblast Activation Protein (FAP), which is highly expressed on cancer-associated fibroblasts within the tumor microenvironment in many epithelial malignancies, including biliary tract cancers. Ga-68 FAPI PET/CT provides high tumor uptake and improved tumor-to-background contrast, which may enhance detection of primary tumors, nodal disease, and distant metastases. It has demonstrated potential advantages over 18F-FDG PET/CT in sensitivity and diagnostic accuracy for staging and recurrence assessment.

SUMMARY:
The goal of this prospective observational study is to evaluate whether Gallium-68 Fibroblast Activation Protein Inhibitor (FAPI) PET/CT can improve detection, staging, and recurrence assessment in adult patients (≥18 years) with suspected or confirmed biliary tract cancers, including gallbladder cancer, cholangiocarcinoma, and post-treatment suspected recurrence.

The main question(s) this study aims to answer are:

Can FAPI PET/CT provide greater sensitivity, specificity and diagnostic accuracy for primary tumors, nodal disease, and metastatic lesions compared to standard FDG PET/CT?

Does FAPI PET/CT offer additional diagnostic yield that may affect clinical decision-making and staging, potentially reducing need for invasive staging procedures?

Researchers will compare FAPI PET/CT with FDG PET/CT to see if FAPI improves detection of metastatic or recurrent disease, especially peritoneal or liver metastasis and lymph node involvement.

Participants will:

Provide written informed consent.

Undergo FAPI PET/CT imaging (baseline and/or at suspected biochemical or radiologic recurrence).

Have quantitative imaging parameters evaluated (SUVmax, tumor-to-liver ratios, metabolic volume).

May undergo comparison with FDG PET/CT and/or follow-up imaging or histopathology as gold standard.

DETAILED DESCRIPTION:
Biliary tract cancers frequently present at an advanced stage and require accurate staging to guide treatment decisions such as surgery, systemic therapy, or palliative management. Although 18 F-FDG PET/CT is widely used in clinical practice, its diagnostic performance is limited in detecting small primary lesions, nodal metastasis, liver metastasis, and peritoneal carcinomatosis. Gallium-68 Fibroblast Activation Protein Inhibitor (FAPI) PET/CT is a novel imaging technology that targets cancer-associated fibroblasts, which are abundant in the desmoplastic stroma characteristic of biliary tract cancers. Early evidence suggests that FAPI PET/CT may provide improved lesion detectability and tumor-to-background contrast compared to FDG PET/CT.

This prospective observational study will evaluate the clinical utility of Ga-68 FAPI PET/CT for initial staging and suspected recurrence in patients with biliary tract cancers. Diagnostic performance metrics (sensitivity, specificity, PPV, NPV, and semi-quantitative PET parameters such as SUVmax and metabolic volume) will be assessed and compared with FDG PET/CT and/or follow-up imaging or histopathology as the gold standard. The study aims to determine the incremental diagnostic contribution of FAPI PET/CT and its potential impact on clinical decision-making.

Findings from this research may help define the role of FAPI PET/CT as a complementary or alternative imaging modality in staging and restaging of biliary tract cancers and may support future prospective multicenter trials.

ELIGIBILITY:
Inclusion Criteria:

* Suspected biliary tract cancers- iHCC and GBC
* Male and females ≥ 18 years;
* Upfront advanced (suspected T3 ,T4, N1, vascular involvement)
* iGBC (residual, N1)
* Suspected post-treatment recurrence (biochemical or radiological)

Exclusion Criteria:

* Informed consent withdrawal
* Concurrent Malignancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include adult male and female patients (≥18 years) with suspected or confirmed biliary tract cancers, including intrahepatic cholangiocarcinoma (iHCC) and gallbladder cancer (GBC). Eligible participants include individuals with upfront advanced disease (suspected T3/T4 tumors, N1 nodal involvement, or vascular involvement), patients with residual or node-positive incidental gallbladder cancer (iGBC), and those with suspected post-treatment recurrence based on biochemical markers or radiologic evaluation.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of Ga-68 FAPI PET/CT for detection of metastatic or recurrent disease (measured as sensitivity and specificity) | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Shraddha Patkar, Principal Investigator — Tata Memorial Hospital
Locations (1):
- Dr.Shraddha Patkar, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pang Y, Zhao L, Luo Z, Hao B, Wu H, Lin Q, Sun L, Chen H. Comparison of 68Ga-FAPI and 18F-FDG Uptake in Gastric, Duodenal, and Colorectal Cancers. Radiology. 2021 Feb;298(2):393-402. doi: 10.1148/radiol.2020203275. Epub 2020 Dec 1. PMID 33258746
- [Background] Chang MC, Chen JH, Liang JA, Huang WS, Cheng KY, Kao CH. PET or PET/CT for detection of peritoneal carcinomatosis: a meta-analysis. Clin Nucl Med. 2013 Aug;38(8):623-9. doi: 10.1097/RLU.0b013e318299609f. PMID 23797225
- [Background] Kim SJ, Lee SW. Diagnostic accuracy of 18F-FDG PET/CT for detection of peritoneal carcinomatosis; a systematic review and meta-analysis. Br J Radiol. 2018 Jan;91(1081):20170519. doi: 10.1259/bjr.20170519. Epub 2017 Nov 21. PMID 29099613
- [Background] Zhao L, Pang Y, Luo Z, Fu K, Yang T, Zhao L, Sun L, Wu H, Lin Q, Chen H. Role of [68Ga]Ga-DOTA-FAPI-04 PET/CT in the evaluation of peritoneal carcinomatosis and comparison with [18F]-FDG PET/CT. Eur J Nucl Med Mol Imaging. 2021 Jun;48(6):1944-1955. doi: 10.1007/s00259-020-05146-6. Epub 2021 Jan 7. PMID 33415432
- [Background] Lan L, Zhang S, Xu T, Liu H, Wang W, Feng Y, Wang L, Chen Y, Qiu L. Prospective Comparison of 68Ga-FAPI versus 18F-FDG PET/CT for Tumor Staging in Biliary Tract Cancers. Radiology. 2022 Sep;304(3):648-657. doi: 10.1148/radiol.213118. Epub 2022 May 17. PMID 35579524
- [Background] Loktev A, Lindner T, Burger EM, Altmann A, Giesel F, Kratochwil C, Debus J, Marme F, Jager D, Mier W, Haberkorn U. Development of Fibroblast Activation Protein-Targeted Radiotracers with Improved Tumor Retention. J Nucl Med. 2019 Oct;60(10):1421-1429. doi: 10.2967/jnumed.118.224469. Epub 2019 Mar 8. PMID 30850501
- [Background] Lindner T, Loktev A, Altmann A, Giesel F, Kratochwil C, Debus J, Jager D, Mier W, Haberkorn U. Development of Quinoline-Based Theranostic Ligands for the Targeting of Fibroblast Activation Protein. J Nucl Med. 2018 Sep;59(9):1415-1422. doi: 10.2967/jnumed.118.210443. Epub 2018 Apr 6. PMID 29626119
- [Background] Goere D, Wagholikar GD, Pessaux P, Carrere N, Sibert A, Vilgrain V, Sauvanet A, Belghiti J. Utility of staging laparoscopy in subsets of biliary cancers : laparoscopy is a powerful diagnostic tool in patients with intrahepatic and gallbladder carcinoma. Surg Endosc. 2006 May;20(5):721-5. doi: 10.1007/s00464-005-0583-x. Epub 2006 Feb 27. PMID 16508808
- [Background] Agarwal AK, Kalayarasan R, Javed A, Gupta N, Nag HH. The role of staging laparoscopy in primary gall bladder cancer--an analysis of 409 patients: a prospective study to evaluate the role of staging laparoscopy in the management of gallbladder cancer. Ann Surg. 2013 Aug;258(2):318-23. doi: 10.1097/SLA.0b013e318271497e. PMID 23059504
- [Background] Petrowsky H, Wildbrett P, Husarik DB, Hany TF, Tam S, Jochum W, Clavien PA. Impact of integrated positron emission tomography and computed tomography on staging and management of gallbladder cancer and cholangiocarcinoma. J Hepatol. 2006 Jul;45(1):43-50. doi: 10.1016/j.jhep.2006.03.009. Epub 2006 Apr 19. PMID 16690156
- [Background] Lamarca A, Barriuso J, Chander A, McNamara MG, Hubner RA, OReilly D, Manoharan P, Valle JW. 18F-fluorodeoxyglucose positron emission tomography (18FDG-PET) for patients with biliary tract cancer: Systematic review and meta-analysis. J Hepatol. 2019 Jul;71(1):115-129. doi: 10.1016/j.jhep.2019.01.038. Epub 2019 Feb 21. PMID 30797051
- [Background] Rodriguez-Fernandez A, Gomez-Rio M, Medina-Benitez A, Moral JV, Ramos-Font C, Ramia-Angel JM, Llamas-Elvira JM, Ferron-Orihuela JA, Lardelli-Claret P. Application of modern imaging methods in diagnosis of gallbladder cancer. J Surg Oncol. 2006 Jun 15;93(8):650-64. doi: 10.1002/jso.20533. PMID 16724342
- [Background] Bedmutha AS, Agrawal A, Rangarajan V, Goel M, Patkar S, Puranik AD, Ramadwar M, Purandare NC, Shah S, Choudhury S. Diagnostic performance of F-18 FDG PET/CT in recurrent adenocarcinoma gallbladder and its impact on post-recurrence survival. Jpn J Radiol. 2023 Feb;41(2):201-208. doi: 10.1007/s11604-022-01340-8. Epub 2022 Sep 19. PMID 36121626
- [Background] Goel M, Tamhankar A, Rangarajan V, Patkar S, Ramadwar M, Shrikhande SV. Role of PET CT scan in redefining treatment of incidental gall bladder carcinoma. J Surg Oncol. 2016 May;113(6):652-8. doi: 10.1002/jso.24198. Epub 2016 Feb 5. PMID 26847023
- [Background] Kang Y, Lee JM, Kim SH, Han JK, Choi BI. Intrahepatic mass-forming cholangiocarcinoma: enhancement patterns on gadoxetic acid-enhanced MR images. Radiology. 2012 Sep;264(3):751-60. doi: 10.1148/radiol.12112308. Epub 2012 Jul 12. PMID 22798225
- [Background] Lim JH. Cholangiocarcinoma: morphologic classification according to growth pattern and imaging findings. AJR Am J Roentgenol. 2003 Sep;181(3):819-27. doi: 10.2214/ajr.181.3.1810819. No abstract available. PMID 12933488
- [Background] STEINER JW, CARRUTHERS JS. Studies on the fine structure of proliferated bile ductules. II. Changes of the ductule-connective tissue envelope relationship. Can Med Assoc J. 1961 Dec 9;85(24):1275-87. No abstract available. PMID 13916730
- [Background] CARRUTHERS JS, KALIFAT SR, STEINER JW. The ductular cell reaction of rat liver in extrahepatic cholestasis. II. The proliferation of connective tissue. Exp Mol Pathol. 1962 Aug;1:377-96. doi: 10.1016/0014-4800(62)90032-1. No abstract available. PMID 13876901
- [Background] Hu K, Li J, Wang L, Huang Y, Li L, Ye S, Han Y, Huang S, Wu H, Su J, Tang G. Preclinical evaluation and pilot clinical study of [18F]AlF-labeled FAPI-tracer for PET imaging of cancer associated fibroblasts. Acta Pharm Sin B. 2022 Feb;12(2):867-875. doi: 10.1016/j.apsb.2021.09.032. Epub 2021 Oct 15. PMID 35256951
- [Background] Hirmas N, Hamacher R, Sraieb M, Ingenwerth M, Kessler L, Pabst KM, Barbato F, Lueckerath K, Kasper S, Nader M, Schildhaus HU, Kesch C, von Tresckow B, Hanoun C, Hautzel H, Aigner C, Glas M, Stuschke M, Kummel S, Harter P, Lugnier C, Uhl W, Niedergethmann M, Hadaschik B, Grunwald V, Siveke JT, Herrmann K, Fendler WP. Fibroblast-Activation Protein PET and Histopathology in a Single-Center Database of 324 Patients and 21 Tumor Entities. J Nucl Med. 2023 May;64(5):711-716. doi: 10.2967/jnumed.122.264689. Epub 2022 Dec 29. PMID 36581374
- [Background] Mona CE, Benz MR, Hikmat F, Grogan TR, Lueckerath K, Razmaria A, Riahi R, Slavik R, Girgis MD, Carlucci G, Kelly KA, French SW, Czernin J, Dawson DW, Calais J. Correlation of 68Ga-FAPi-46 PET Biodistribution with FAP Expression by Immunohistochemistry in Patients with Solid Cancers: Interim Analysis of a Prospective Translational Exploratory Study. J Nucl Med. 2022 Jul;63(7):1021-1026. doi: 10.2967/jnumed.121.262426. Epub 2021 Nov 5. PMID 34740953
- [Background] Kratochwil C, Flechsig P, Lindner T, Abderrahim L, Altmann A, Mier W, Adeberg S, Rathke H, Rohrich M, Winter H, Plinkert PK, Marme F, Lang M, Kauczor HU, Jager D, Debus J, Haberkorn U, Giesel FL. 68Ga-FAPI PET/CT: Tracer Uptake in 28 Different Kinds of Cancer. J Nucl Med. 2019 Jun;60(6):801-805. doi: 10.2967/jnumed.119.227967. Epub 2019 Apr 6. PMID 30954939
- [Background] Baum RP, Schuchardt C, Singh A, Chantadisai M, Robiller FC, Zhang J, Mueller D, Eismant A, Almaguel F, Zboralski D, Osterkamp F, Hoehne A, Reineke U, Smerling C, Kulkarni HR. Feasibility, Biodistribution, and Preliminary Dosimetry in Peptide-Targeted Radionuclide Therapy of Diverse Adenocarcinomas Using 177Lu-FAP-2286: First-in-Humans Results. J Nucl Med. 2022 Mar;63(3):415-423. doi: 10.2967/jnumed.120.259192. Epub 2021 Jun 24. PMID 34168013
- [Background] Zhao L, Niu B, Fang J, Pang Y, Li S, Xie C, Sun L, Zhang X, Guo Z, Lin Q, Chen H. Synthesis, Preclinical Evaluation, and a Pilot Clinical PET Imaging Study of 68Ga-Labeled FAPI Dimer. J Nucl Med. 2022 Jun;63(6):862-868. doi: 10.2967/jnumed.121.263016. Epub 2021 Sep 23. PMID 34556528
- [Background] Poplawski SE, Lai JH, Li Y, Jin Z, Liu Y, Wu W, Wu Y, Zhou Y, Sudmeier JL, Sanford DG, Bachovchin WW. Identification of selective and potent inhibitors of fibroblast activation protein and prolyl oligopeptidase. J Med Chem. 2013 May 9;56(9):3467-77. doi: 10.1021/jm400351a. Epub 2013 Apr 29. PMID 23594271
- [Background] Ishii G, Ochiai A, Neri S. Phenotypic and functional heterogeneity of cancer-associated fibroblast within the tumor microenvironment. Adv Drug Deliv Rev. 2016 Apr 1;99(Pt B):186-196. doi: 10.1016/j.addr.2015.07.007. Epub 2015 Aug 14. PMID 26278673
- [Background] Liao Z, Tan ZW, Zhu P, Tan NS. Cancer-associated fibroblasts in tumor microenvironment - Accomplices in tumor malignancy. Cell Immunol. 2019 Sep;343:103729. doi: 10.1016/j.cellimm.2017.12.003. Epub 2018 Feb 13. PMID 29397066
- [Background] Jacob M, Chang L, Pure E. Fibroblast activation protein in remodeling tissues. Curr Mol Med. 2012 Dec;12(10):1220-43. doi: 10.2174/156652412803833607. PMID 22834826
- [Background] Kinnman N, Francoz C, Barbu V, Wendum D, Rey C, Hultcrantz R, Poupon R, Housset C. The myofibroblastic conversion of peribiliary fibrogenic cells distinct from hepatic stellate cells is stimulated by platelet-derived growth factor during liver fibrogenesis. Lab Invest. 2003 Feb;83(2):163-73. doi: 10.1097/01.lab.0000054178.01162.e4. PMID 12594232
- [Background] Beaussier M, Wendum D, Schiffer E, Dumont S, Rey C, Lienhart A, Housset C. Prominent contribution of portal mesenchymal cells to liver fibrosis in ischemic and obstructive cholestatic injuries. Lab Invest. 2007 Mar;87(3):292-303. doi: 10.1038/labinvest.3700513. Epub 2007 Jan 29. PMID 17260005
- [Background] Apte MV, Haber PS, Applegate TL, Norton ID, McCaughan GW, Korsten MA, Pirola RC, Wilson JS. Periacinar stellate shaped cells in rat pancreas: identification, isolation, and culture. Gut. 1998 Jul;43(1):128-33. doi: 10.1136/gut.43.1.128. PMID 9771417
- [Background] Hasegawa T, Yashiro M, Nishii T, Matsuoka J, Fuyuhiro Y, Morisaki T, Fukuoka T, Shimizu K, Shimizu T, Miwa A, Hirakawa K. Cancer-associated fibroblasts might sustain the stemness of scirrhous gastric cancer cells via transforming growth factor-beta signaling. Int J Cancer. 2014 Apr 15;134(8):1785-95. doi: 10.1002/ijc.28520. Epub 2013 Oct 24. PMID 24155219
- [Background] Landskron G, De la Fuente M, Thuwajit P, Thuwajit C, Hermoso MA. Chronic inflammation and cytokines in the tumor microenvironment. J Immunol Res. 2014;2014:149185. doi: 10.1155/2014/149185. Epub 2014 May 13. PMID 24901008
- [Background] Kubo S, Takemura S, Tanaka S, Shinkawa H, Kinoshita M, Hamano G, Ito T, Koda M, Aota T. Occupational cholangiocarcinoma caused by exposure to 1,2-dichloropropane and/or dichloromethane. Ann Gastroenterol Surg. 2017 Nov 17;2(2):99-105. doi: 10.1002/ags3.12051. eCollection 2018 Mar. PMID 29863124
- [Background] Kubo S, Takemura S, Tanaka S, Shinkawa H, Kinoshita M, Hamano G, Ito T, Koda M, Aota T, Yamamoto T, Terajima H, Tachiyama G, Yamada T, Nakamori S, Arimoto A, Fujikawa M, Tomimaru Y, Sugawara Y, Nakagawa K, Unno M, Mizuguchi T, Takenaka K, Kimura K, Shirabe K, Saiura A, Uesaka K, Taniguchi H, Fukuda A, Chong JM, Kuwae Y, Ohsawa M, Sato Y, Nakanuma Y. Outcomes after resection of occupational cholangiocarcinoma. J Hepatobiliary Pancreat Sci. 2016 Sep;23(9):556-64. doi: 10.1002/jhbp.373. Epub 2016 Aug 1. PMID 27363864
- [Background] Ham IH, Lee D, Hur H. Role of Cancer-Associated Fibroblast in Gastric Cancer Progression and Resistance to Treatments. J Oncol. 2019 Jun 9;2019:6270784. doi: 10.1155/2019/6270784. eCollection 2019. PMID 31281359
- [Background] Hanahan D, Coussens LM. Accessories to the crime: functions of cells recruited to the tumor microenvironment. Cancer Cell. 2012 Mar 20;21(3):309-22. doi: 10.1016/j.ccr.2012.02.022. PMID 22439926
- [Background] Ohira M, Kobayashi T, Hashimoto M, Tazawa H, Abe T, Oshita A, Kohashi T, Irei T, Oishi K, Ohdan H; Hiroshima Surgical study group of Clinical Oncology (HiSCO). Prognostic factors in patients with recurrent intrahepatic cholangiocarcinoma after curative resection: A retrospective cohort study. Int J Surg. 2018 Jun;54(Pt A):156-162. doi: 10.1016/j.ijsu.2018.04.058. Epub 2018 May 3. PMID 29730072
- [Background] Zheng J, Cai J, Tao L, Kirih MA, Shen Z, Xu J, Liang X. Comparison on the efficacy and prognosis of different strategies for intrahepatic recurrent hepatocellular carcinoma: A systematic review and Bayesian network meta-analysis. Int J Surg. 2020 Nov;83:196-204. doi: 10.1016/j.ijsu.2020.09.031. Epub 2020 Sep 25. PMID 32980518
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338